CLINICAL TRIAL: NCT00574405
Title: Preservation of Pancreatic Beta Cell Function Through Insulin Pump Therapy
Acronym: ktpump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29256; CUMG - 090104KT
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
Keywords: Insulin pump; Beta cell
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin; Insulin Glargine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): MDI = 3-4+ insulin injections/day, using split-mix NPH insulin + regular insulin or Lantus + Novolog® (or Humalog®).
  Interventions: Drug: MDI (split-mix NPH insulin + regular insulin or Lantus + Novolog® [or Humalog®])
- 2 (Experimental): CSII (insulin pump), using Animas Corporation insulin pump, model IR 1200.
  Interventions: Device: CSII (Animas Corporation insulin pump, model IR 1200)

INTERVENTIONS:
Drug: MDI (split-mix NPH insulin + regular insulin or Lantus + Novolog® [or Humalog®]) — MDI = 3-4+ insulin injections/day, using NPH + regular insulin or Lantus + insulin lispro; 12 month treatment duration.
  Other Names: Novolog® or Humalog®
  Arms: 1
Device: CSII (Animas Corporation insulin pump, model IR 1200) — CSII (insulin pump), using Animas Corporation insulin pump, model IR 1200.
  Other Names: Animas Corporation insulin pump, model IR 1200
  Arms: 2

SUMMARY:
Type I diabetes (T1DM) is the second most common chronic illness effecting children in the USA. Worldwide, Type I diabetes is increasing in incidence, and its underlying etiology remains elusive. Nevertheless, recent data supports the notion that early and intensive management of Type I diabetes can 1) decrease long-term complications of diabetes; and 2) may significantly improve beta cell function and insulin secretion over ensuing years. To this end, we propose using insulin pump therapy to preserve and/or enhance residual endogenous B-cell secretory capacity among patients with newly diagnosed Type 1 DM. Furthermore, we anticipate that early use of an insulin pump will improve glycemic control beyond that achieved with standard multiple daily injection (MDI) therapy, and will be well-tolerated by the patient. These data will provide important pilot information to explore the potential role of intensive insulin pump therapy in the treatment of children newly diagnosed with Type I diabetes. The specific aim of this study is to test the following hypothesis: Early use of insulin pump therapy is effective in preserving or enhancing residual endogenous pancreatic B-cell secretory capacity among patients with newly diagnosed T1DM: Moreover, early use of an insulin pump will improve glycemic control beyond that achieved with standard multiple injection therapy, and will be well-tolerated by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Medical history and clinical presentation consistent with the diagnosis of Type 1 DM.
* Age: 8-18 years

Exclusion Criteria:

* Clinical presentation consistent with Type 2 DM.
* History of other chronic systemic inflammatory or autoimmune disease or other severe medical conditions.
* Concurrent pregnancy.
* Participation in other research protocols or use of other investigational agents within 30 days of enrollment.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Thrailkill, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital/Research Institute, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 children with T1D were screened between 04/05-02/09; 64 declined to participate; 16 did not meet inclusion/exclusion criteria. 24 subjects (12 per group) were enrolled. 1 subject in each group withdrew after initial randomization. Of the remaining 22, 1 completed the 9-mo visit, 1 completed the 6-mo visit, and 1 completed the 1-mo visit.
Pre-assignment Details: One subject in each group withdrew from further participation after initial randomization, possibly because of dissatisfaction with the assigned mode of treatment.
Groups:
- Multiple Daily Injection Therapy: Multiple daily injection therapy, using split-mix NPH insulin + regular insulin or Lantus + Novolog® (or Humalog®) started at the time of diagnosis of Type 1 diabetes in patient 8-18 years of age and monitored for 12 months after diagnosis.
- Insulin Pump Therapy, Started at Diagnosis.: Continuous subcutaneous infusion therapy (insulin pump therapy), using Animas Corporation insulin pump, model IR 1200, started within 1 month of diagnosis with Type 1 diabetes, in patients 8-18 years of age, and monitored for 12 months after diagnosis.
Period: Overall Study
Arm/Group | Multiple Daily Injection Therapy | Insulin Pump Therapy, Started at Diagnosis.
Started | 12 | 12
Completed | 9 | 10
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Daily Injection Therapy | Insulin Pump Therapy, Started at Diagnosis. | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (2.5) | 12.1 (3.6) | 12.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Mixed-meal-stimulated Peak C-peptide Value (Via Mixed-meal Tolerance Test) After 12 Months of Insulin Pump Therapy, Compared With MDI.
Time Frame: 12 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Multiple Daily Injection Therapy | Insulin Pump Therapy, Started at Diagnosis.
Number analyzed (Participants) | 9 | 10
ng/mL | 1.8 (1.4) | 3.1 (2.2)

2. Secondary Outcome: Changes in Glycemic Control, as Assessed by the Change in Hemoglobin A1c and Variations in Daily Blood Glucose Measurements (Fasting BG and CGMS) From Day 1 of Treatment to Month 12 of Treatment.
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Daily Insulin Requirements Over Time
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Frequency of Adverse Glycemic Consequences, i.e., Frequency of Hypoglycemia, Severe Hyperglycemia or Ketosis.
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Patient Satisfaction With Mode of Therapy and Patient Compliance With Treatment Recommendations.
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Multiple Daily Injection Therapy | Insulin Pump Therapy, Started at Diagnosis.
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 10/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Daily Injection Therapy (N=12) | Insulin Pump Therapy, Started at Diagnosis. (N=12)
Hospitilized for treatment of Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Subject was hospitilized in a local hospital for initial treatment of symptoms of a urinary tract infection; discharged home on oral antibiotics, in good condition. Patient had a history of recurrent UTIs, prior to study enrollment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Daily Injection Therapy (N=12) | Insulin Pump Therapy, Started at Diagnosis. (N=12)
Abdominal pain/constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pump malfunction (Investigations) | 0 (0) | 4 (4)
Infections (Infections and infestations) | 7 (13) | 5 (10)
Injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Vision change (Eye disorders) | 2 (3) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Post hoc analysis demonstrated that the study design was weakened by an underestimation of the sample size per group needed to determine a statistically significant result for our primary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less